CLINICAL TRIAL: NCT05189886
Title: Transcatheter Aortic Valve Replacement (TAVR) Double Balloon Valvuloplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Community Memorial Health System (Other)
Responsible Party: Principal Investigator, Jennifer Wan, Attending Physician, Community Memorial Health System
Other Study IDs: 2021-HSR013
Record Dates: First submitted 2021-11-22; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; Balloon Valvuloplasty
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: The prospective phase will enroll patients planning to undergo TAVR, at the discretion of Drs. Wan and Fatemi, and if they meet all of the inclusion criteria and none of the exclusion criteria. All patients who provide consent will undergo the TAVR procedure where the valve will be double inflated. Echocardiogram results and procedure details will be collected as data. At the patient's 30-day follow-up clinic visit, as per standard of care, they will be re-evaluated with an echocardiogram. Details from that follow-up visit and the echocardiogram results will be collected as data. Prospective enrollment will begin upon IRB approval and we plan to continue enrollment until December 31, 2023, or once 200 participants are reached, whichever comes first.
  Interventions: Procedure: Double Balloon Valvuloplasty in TAVR
- Retrospective: The retrospective phase will collect data from previous TAVR procedures completed between February 2019 and October 1, 2021. Data from up to 200 patient charts will be collected using the Society of Thoracic Surgeons/American College of Cardiology that is maintained by the CMH Cardiology Department. The population will be de-identified as the purpose is to obtain descriptive information from the medical records to utilize for propensity match scoring.

INTERVENTIONS:
Procedure: Double Balloon Valvuloplasty in TAVR — The prospective phase will enroll patients planning to undergo TAVR, at the discretion of Drs. Wan and Fatemi, and if they meet all of the inclusion criteria and none of the exclusion criteria. All patients who provide consent will undergo the TAVR procedure where the valve will be double inflated. Echocardiogram results and procedure details will be collected as data. At the patient's 30-day follow-up clinic visit, as per standard of care, they will be re-evaluated with an echocardiogram. Details from that follow-up visit and the echocardiogram results will be collected as data. Prospective enrollment will begin upon IRB approval and we plan to continue enrollment until December 31, 2023, or once 200 participants are reached, whichever comes first.
  Groups: Prospective

SUMMARY:
In this study, the investigators evaluate whether routine double inflation of the valve could have a lasting impact. The investigators hypothesize that a routine second reinflation of the balloon, or "double tap", will improve flow across the valve when compared to a single inflation. The investigators hypothesize that "double tap" (1) will decrease mean gradient between first and second inflation during the procedure, (2) will decrease mean gradient on immediate post procedure and 30 day postprocedure echocardiograms when compared to mean gradient gradient after single inflation. Less obstruction indicated by lower mean gradient early after deployment may translate to improved 5 and 10 year outcomes. Furthermore, the investigators hypothesize that this small change in technique will have no effect on procedure time or complications and the change will not result in any increase in perioperative vascular complications, or new permanent pacemaker insertion.

The primary objective of this study is to determine if double valve inflation during a TAVR procedure improves valve area and mean gradients as measured by echocardiogram immediately following the procedure and at 30 days follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Diagnosis of severe native valve aortic stenosis
3. Meets the standard of care indications to undergo TAVR procedure (aortic valve area <1.0 cm2 or mean pressure gradient >40 mmHg or peak velocity >4.0 m/s or aortic valve area index <0.6).
4. Provided informed consent.

Exclusion Criteria:

1. History of prior aortic valve replacement
2. Pre-existing moderate to severe aortic regurgitation
3. Lacking pre-procedure echocardiogram
4. Patients planning to undergo multiple valve replacements simultaneously
5. Intraoperative arrhythmia
6. Intraoperative hemodynamic instability
7. Intraoperative complication during initial inflation (such as: aortic dissection, coronary artery occlusion, coronary artery dissection)
8. At the discretion of the principal investigator, any reason that the potential subject may be unfit for participation, such as frailty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient with moderate to severe aortic regurgitation requiring replacement of his/her aortic valve.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Valve area | Immediately following the procedure
  Valve area as measured by echocardiogram
Valve area | At 30 days follow up
  Valve area as measured by echocardiogram
Mean gradient | Immediately following the procedure
  Mean gradient as measured by echocardiogram
Mean gradient | At 30 days follow up
  Mean gradient as measured by echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wan, MD, Principal Investigator — Community Memorial HealthCenter
Locations (1):
- Community Memorial Hospital, Ventura, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT05189886/ICF_000.pdf